CLINICAL TRIAL: NCT05849246
Title: Open-label, Phase 2 Study of Tusamitamab Ravtansine (IBI126) Combined With Sintilimab and Tusamitamab Ravtansine (IBI126) Combined With Sintilimab Plus Platinum-based Chemotherapy and Pemetrexed in Subjects With CEACAM5 Positive Expression Advanced/Metastatic Non-squamous Non-small-cell Lung Cancer (NSQ NSCLC)
Brief Title: The Study of Tusamitamab Ravtansine (IBI126) Combined With Sintilimab and Tusamitamab Ravtansine (IBI126) Combined With Sintilimab Plus Platinum-based Chemotherapy and Pemetrexed in Subjects With CEACAM5 Positive Expression Advanced/Metastatic Non-squamous Non-small-cell Lung Cancer (NSQ NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: strategy terminates development, the decision is not due to any safety-related issues
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI126A201
Record Dates: First submitted 2023-04-17; First posted 2023-05-08 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Non-squamous Non-small-cell Lung Cancer
Keywords: CEACAM5

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tusamitamab ravtansine + sintilimab (Experimental): Sintilimab dose will be administered intravenously prior to intravenous administration of tusamitamab ravtansine dose every 3 weeks.
  Interventions: Drug: Tusamitamab ravtansine+Sintilimab
- Tusamitamab ravtansine + Sintilimab + carboplatin/ cisplatin + pemetrexed (Experimental): Sintilimab dose will be administered intravenously prior to intravenous adminstration of tusamitamab ravtansine dose every 3 weeks. Pemetrexed will be infused over 10 minutes after tusamitamab ravtansine infusion on Day 1 and then Q3W. Carboplatin / cisplatin will be infused over 15 to 60 minutes immediately after pemetrexed infusion on Day 1 and Q3W for the first 4 cycles.
  Interventions: Drug: Tusamitamab ravtansine+Sintilimab+Carboplatin or Cisplatin+Pemetrexed
- Sintilimab + carboplatin/ cisplatin + pemetrexed (Placebo Comparator): Pemetrexed will be infused over 10 minutes after Sintilimab infusion on Day 1 and then Q3W. Carboplatin/ cisplatin will be infused over 15 to 60 minutes immediately after pemetrexed infusion on Day 1 and Q3W for the first 4 cycles.
  Interventions: Drug: Sintilimab+Carboplatin or Cisplatin+Pemetrexed

INTERVENTIONS:
Drug: Tusamitamab ravtansine+Sintilimab+Carboplatin or Cisplatin+Pemetrexed — Pharmaceutical form: Concentrate for solution for infusion Route of administration: Intravenous.
  Other Name: Tusamitamab ravtansine. Other Name: Tyvyt®
  Arms: Tusamitamab ravtansine + Sintilimab + carboplatin/ cisplatin + pemetrexed
Drug: Sintilimab+Carboplatin or Cisplatin+Pemetrexed — Pharmaceutical form: Concentrate for solution for infusion Route of administration: Intravenous
  Arms: Sintilimab + carboplatin/ cisplatin + pemetrexed
Drug: Tusamitamab ravtansine+Sintilimab — Pharmaceutical form:Concentrate for solution for infusion Route of administration: Intravenous.
  Other Name: Tusamitamab ravtansine. Other Name: Tyvyt®
  Arms: tusamitamab ravtansine + sintilimab

SUMMARY:
Primary objective：

·To assess the antitumor activity of tusamitamab ravtansine in combination with sintilimab and tusamitamab ravtansine in combination with sintilimab, platinum-based chemotherapy and pemetrexed in the NSQ NSCLC population.

Secondary objectives： To assess the safety and tolerability of tusamitamab ravtansine in combination with sintilimab and tusamitamab ravtansine in combination with sintilimab, platinum-based chemotherapy and pemetrexed in the NSQ NSCLC population.

To assess the pharmacokinetic (PK) characteristic of tusamitamab ravtansine in combination with sintilimab and tusamitamab ravtansine in combination with sintilimab, platinum-based chemotherapy and pemetrexed in the NSQ NSCLC population.

DETAILED DESCRIPTION:
The expected duration of the study intervention for participants may vary based on progression date; median expected duration of study per participant is estimated 10 months (up to 1 month for screening, a median of 6 months for treatment, and a median of 3 months for end-of-treatment assessments and safety follow-up visit).

ELIGIBILITY:
Inclusion criteria apply:

I1. Age ≥ 18 years and < 75 years males of females.

I2. Histologically- or cytologically-confirmed diagnosis of advanced or metastatic NSQ NSCLC with no EGFR sensitizing mutation, BRAF mutation or ALK/ROS alterations.

I3. No prior systemic therapy for the treatment of advanced or metastatic disease.

I4. Expression of CEACAM5 as demonstrated prospectively by a centrally assessed IHC assay with ≥ 2+ in intensity involving at least 1% of the tumor cell population in archival tumor sample (or if not, available fresh biopsy sample will be collected if considered an acceptable risk by the treating physician).

I5. Adequate hematologic/liver/renal/coagulation function.

I6. Life expectancy exceeds 3 months.

I7. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion criteria:

E1. Hstologically or cytologically confirmed mixed NSCLC with small-cell or prodominant squamous carcinoma components.

E2. Unstable brain metastases and history of leptomeningeal disease.

E3. Significant concomitant illness, including any severe medical conditions that, in the opinion of the investigator or sponsor, would impair the subject's participation in the study or interpretation of the results.

E4. History within the last 3 years of an invasive malignancy other than the one treated in this study, with the exception of resected/ablated basal or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix, or other local tumors considered cured by local treatment.

E5. History of known acquired immunodeficiency syndrome (AIDS) related illnesses or known HIV disease requiring antiretroviral treatment, or active hepatitis A, B (defined as either positive HBsAg or positive hepatitis B viral DNA test above the lower limit of detection of the assay), or C (defined as a known positive hepatitis C antibody result and known quantitative HCV RNA results greater than the lower limits of detection of the assay) infection.

E6. History of active autoimmune disease that has required systemic treatment in the past 2 years.

E7. Non-resolution of any prior treatment-related toxicity to < Grade 2 according to NCI CTCAE V5.0, with the exception of alopecia, vitiligo, or active thyroiditis controlled with hormone-replacement therapy.

E8. Unresolved corneal disorder or any previous corneal disorder considered by an ophthalmologist to predict higher risk of drug-induced keratopathy. The use of contact lenses is not permitted. Patients using contact lenses who are not willing to stop wearing them for the duration of the study intervention are excluded.

E9. Received traditional Chinese medicine with anti-tumor indications within 2 weeks prior the first administration, or received immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use for pleural effusion control) within 2 weeks prior administration.

E10. Have received prior systemic therapy for advanced/metastatic NSCLC.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) per RECIST 1.1 by investigators. | 3 years
  ORR is defined as proportion of participants who have a confirmed complete

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) and laboratory abnormalities | 3 years
  TEAEs, SAEs and laboratory abnormalities according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).
Pharmacokinetic concentrations of tusamitamab ravtansine (IBI126) | 3 years
Duration of Response (DoR) | 3 years
  DoR is defined the time when subject reaches complete or partial response for the first time to the progression of the disease.
Progression-free Survival (PFS) | 3 years
Time to Response (TTR) | 3 years
Disease Control Rate (DCR) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China